CLINICAL TRIAL: NCT05288582
Title: Tear Lipid Layer Thickness Assessments With Perfluorohexyloctane Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jennifer Fogt, PI, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021H0436
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All participants will be given the eye drop and will have their tear lipid examined before and after use of the drop.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perfluorohexyloctane eye drop (Other): Participants will have their tear lipid layer assessed. They will then have the eye drop instilled and will have an additional assessment of the tear lipid layer within 5 minutes of instillation of the the drop, and again 15 minutes after instillation.
  Interventions: Device: NovaTears

INTERVENTIONS:
Device: NovaTears — Over-the-counter eye drop

SUMMARY:
The purpose of this study is to explore the tear lipid layer quantitatively and qualitatively before and after use of a perflurohexyloctane eye drop (NovaTears)

DETAILED DESCRIPTION:
The tear lipid layer will be studied before and after the use of an over-the-counter eye drop (NovaTears, Novaliq GmbH, Heidelberg, Germany) using a Stroboscopic Video Color Microscope, which is non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* • Age - at least 30 years

  * Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI)
  * Ability to give informed consent
  * Willing to spend time for the study; approximately one hour for a screening visit and 45 minutes for a data collection visit.
  * Either gender
  * Any racial or ethnic origin
  * tear lipid thickness ≤ 75 nm

Exclusion Criteria:

* Active ocular inflammation
* Use of any ocular prescription medication (such as but not limited to, glaucoma medications, anti-inflammatory eye drops and Restasis or Xiidra) used within 14 days of the screening visit or started prior to the measurement visit(s).
* Currently having punctal plugs inserted in lacrimal puncta
* Current eye disease, infection or inflammation that affects the surface of the eye such as, but not limited to moderate or greater blepharitis and ocular allergy. Clinically significant (active treatment) of blepharitis, Sjogren's disease or other systemic disease that could influence MGD, corneal, conjunctival, or eyelid abnormalities that could influence lipid layer thickness, conjunctivitis of any cause, ocular infection or systemic medication such as diuretics, SSRIs, that could influence tear secretion, or sensitivity to any of the ingredient in the eye drop being tested,
* Past eye surgery, such as, but not limited to, refractive surgery. Subjects who have had cataract removal surgery more than one year ago may be considered as potential subjects.
* Female subjects may not be pregnant or lactating. (Subject will be asked to self-report these conditions.)
* Infectious diseases (for example, hepatitis, tuberculosis) or an immuno-suppressive disease (for example, HIV). (Subjects will be asked to self-report these conditions.)
* Inability to complete the screening and examination
* Inability to provide analyzable data. For example, subjects who cannot keep their eye open during the entire measurement interval (due to early blinking) or provide a readable eye image (due to eyelid laxity) or cannot sit still for 1 minute.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Tear lipid layer thickness | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fogt, OD MS, Principal Investigator — OSU College of Optometry
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No